CLINICAL TRIAL: NCT05666674
Title: Software-based Modification of Hand Tremors in XR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: NeuroStorm, Inc (Industry)
Collaborators: stoPD.org (Unknown)
Responsible Party: Principal Investigator, eMalick G. Njie, Chief Scientist, NeuroStorm, Inc
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0224506734
Record Dates: First submitted 2022-12-18; First posted 2022-12-28 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Tremor
MeSH Terms: conditions — Tremor

STUDY DESIGN:
Intervention Model Description: The trial will be composed of two arms: an experimental group with VR with activated Tremor Stabilization Algorithms (TSA-ON). And an active comparator group that is exposed to VR without Tremor Stabilization Algorithms (TSA-OFF control). In both arms, study subjects will be immersed in a stock VR testing environment and will perform a tremor eliciting PTT test.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TSA-ON (Experimental): The trial will be composed of two arms: an experimental group with VR with activated Tremor Stabilization Algorithms (TSA-ON). And an active comparator group that is exposed to VR without Tremor Stabilization Algorithms (TSA-OFF control). In both arms, study subjects will be immersed in a stock VR testing environment and will perform a tremor eliciting PTT test.
  Interventions: Other: TSA algorithms
- TSF-OFF control (Active Comparator): The trial will be composed of two arms: an experimental group with VR with activated Tremor Stabilization Algorithms (TSA-ON). And an active comparator group that is exposed to VR without Tremor Stabilization Algorithms (TSA-OFF control). In both arms, study subjects will be immersed in a stock VR testing environment and will perform a tremor eliciting PTT test.
  Interventions: Other: TSA algorithms

INTERVENTIONS:
Other: TSA algorithms — Our study will be composed of an experimental and an active comparator (i.e., control) arm. Both arms will perform a postural tremor test (PTT) to elicit parkinsonian tremors. The PTT is where subjects stabilize their backs against a wall and position their hands in the air against gravity for two minutes. The experimental arm will receive VR plus activated Tremor Stabilization Algorithms (TSA-ON) while the active comparator arm will receive VR only (TSA-OFF). Thus, subjects in the experimental arm will not see their digital arms tremor while those in the active comparator arm will. Our primary outcome is the severity of PTT elicited tremors. Tremors will be recorded by VR motion-capture controllers.

SUMMARY:
The following trial evaluates the effect of Tremor Stabilization Algorithms on involuntary hand tremors suffered by Parkinson's patients. These algorithms will be implemented in Virtual Reality (VR). Approximately 300 study subjects are to be randomized to experimental (VR plus algorithms, i.e., intervention) and active comparator (VR only, i.e., control) study arms. Study subjects will perform a postural tremor test (PTT) to elicit postural parkinsonian tremors. Our primary outcome is whether the intervention modifies tremor severity.

DETAILED DESCRIPTION:
The following trial evaluates the effect of Tremor Stabilization Algorithms on involuntary hand tremors suffered by Parkinson's patients. These algorithms will be implemented in Virtual Reality (VR). Approximately 300 study subjects are to be randomized to experimental (VR plus algorithms, i.e., intervention) and active comparator (VR only, i.e., control) study arms. Study subjects will perform a postural tremor test (PTT) to elicit postural parkinsonian tremors. Our primary outcome is whether the intervention modifies tremor severity. Secondary outcomes include determining whether tremor severity is reduced long-term. These measurements will occur 5 minutes to 30 days post-intervention and will not involve VR. Other secondary outcomes include determining age-of-onset impact on tremor severity, and online self-report surveys for functionality in life in general and in the context of Parkinson's disease. Subjects will perform tremor-recordings on-site. Self-reports will be remote.

ELIGIBILITY:
Inclusion Criteria:

* Candidates eligible for our study will be 35 - 85 years, diagnosed with Parkinson's disease, with no falls within 6 months prior to the study, are able to walk for 5 minutes unassisted, have adequate hearing and vision capabilities, can comply with study requirements, have the ability to fill online questionnaires, and provide written informed consent to participate in the study.

Exclusion Criteria:

* Candidates that are ineligible for our study have visual-perceptual deficits that limit capacity to be in VR, have clinical diagnosis of dementia or other severe cognitive impairment as determined by a Mini-Mental State Examination score (MMSE) of less than 24, or have a history of stroke, traumatic brain injury or other neurological disorders

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Tremor reduction | 1 minute
  Our primary outcome is the severity of PTT elicited tremors. Tremors will be recorded by VR motion-capture controllers. Wavelet transformation of this data will be applied to determine tremor severity in the two study arms.

CONTACTS AND LOCATIONS:
Locations (1):
- NeuroStorm, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided